CLINICAL TRIAL: NCT02945059
Title: Multicentric Prospective Study Assessing the Efficiency of Preoperative Reversible Selective Portal Vein Embolization in Patients Requiring Major Hepatic Resection
Brief Title: Reversible Portal Vein Embolization Before Major Hepatectomy
Acronym: EMBORES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P150953
Record Dates: First submitted 2016-10-17; First posted 2016-10-26 (Estimated); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Liver Regeneration; Reversible Portal Vein Embolization
Keywords: Liver regeneration; portal vein embolization; gelatin powder; liver surgery; hepatectomy

STUDY DESIGN:
Intervention Model Description: Reversible Portal vein embolization (PVE) using curaspon® (Absorbable Gelatin Hemostats)
Masking Description: Single-arm feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Patients will undergo reversible PVE before major hepatic resection.
  Interventions: Procedure: Selective reversible portal vein embolization

INTERVENTIONS:
Procedure: Selective reversible portal vein embolization — Percutaneous access to the portal vein is achieved under general anesthesia with ultrasound or fluoroscopic control. After assessment of portal venous anatomy, embolization of selected portal vein segments is performed using the powdered form of an absorbable gelatin sponge.

SUMMARY:
The aim of this study is to prospectively evaluate the tolerance and efficiency of a new technique of preoperative selective portal vein embolization (PVE) in patients requiring major hepatic resection.

DETAILED DESCRIPTION:
Portal vein embolization (PVE) is used before major hepatectomy to induce hypertrophy of the future liver remnant (FLR). A non-reversible absorbable material is generally used for embolization, as it provides effective, permanent vascular occlusion. Our team has developed a minimally invasive technique of reversible PVE using gelfoam powder. The aim of this study is to assess the tolerance and efficiency of preoperative reversible selective PVE in patients requiring major hepatic resection. We hypothesize that preoperative reversible PVE allows to similarly increase FLR volume in comparison with classical non-reversible PVE in patients requiring major liver resection with limited FLR.

The hypertrophy ratio after classical non-reversible PVE is evaluated in literature as 13%. We estimated the hypertrophy ratio after reversible PVE as 9% in a previous retrospective study.

The aim of this pilot study is to prospectively evaluate the hypertrophy ratio after reversible PVE.

Primary End Point: Hypertrophy ratio of FLR volume / total liver volume between the baseline and after PVE, assessed by computed tomography scan volumetry 4-6 weeks after PVE.

ELIGIBILITY:
Inclusion Criteria:

Patient aged between 18 and 80 years

* Patient requiring major liver resection (at least 3 segments)
* PVE indication decided in a multidisciplinary meeting
* Patients who are able to understand and follow instructions and who are able to participate in the study for the entire period
* Patients must have given their written informed consent to participate in the study after having received adequate previous information and prior to any study-specific procedures
* Patient affiliated to the French National Social Security System

Exclusion Criteria:

* American Score of Anesthesiologist (ASA) > 3
* Extensive Portal vein or hepatic vein thrombosis
* Patient not covered by social security service
* Patient under guardianship
* Patients with a medical disorder, condition, or history of such that would impair the patient's ability to participate or complete this study in the opinion of the investigator.
* Patients who have already had anaphylactic or anaphylactoid reactions during the injection of iodinated contrast medium (edema of Quincke…)
* Patients with an allergy to pork products During the hospitalization and before the PVE
* Severe renal insufficiency (glomerular filtration rate ≤ 30mL/min eg calculated based on the Cockcroft formula).
* Pregnant women, or breast feeding women, or women with childbearing potential not using a combination of condoms and a safe and highly effective contraception method during the participation to the research (hormonal contraception with implants or oral contraceptives, or intrauterine devices).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Hypertrophy ratio of FLR volume / total liver volume between the baseline and after the PVE | 4-6 weeks after portal vein embolization
  Ratio is evaluated by computed tomography scan volumetry 4-6 weeks after portal vein embolization.Volumes will be assessed by one independent blind observer, from anonymized CT scan series. Total, non-embolized (FLR) volume and embolized liver volume (ELV) will be measured.
  The following formulas will be used to calculate percentage of FLR volume:
  * FLR volume prePVE = (FLR prePVE volume / (total liver prePVE volume - tumor volume prePVE)) x 100
  * FLR volume postPVE = (FLR postPVE volume / (total liver postPVE volume - tumor volume postPVE)) x 100
  The following formulas will be used to calculate hypertrophy ratio:
  %FLR volume postPVE - %FLR volume prePVE

SECONDARY OUTCOMES:
Technical feasibility: Percentage of completed PVE | During the procedure of portal vein embolization
  Percutaneous access to the portal vein is achieved under general anesthesia with ultrasound or fluoroscopic control. Venous cartography of the liver is achieved with fluoroscopic control. PVE technique remains unchanged but a mixture of absorbable embolization agent is injected.
  Adverse events will be questioned and documented in the electronic Case Report Form.
Technical feasibility: Percentage of partially completed PVE | During the procedure of portal vein embolization
  Percutaneous access to the portal vein is achieved under general anesthesia with ultrasound or fluoroscopic control. Venous cartography of the liver is achieved with fluoroscopic control. PVE technique remains unchanged but a mixture of absorbable embolization agent is injected.
  Adverse events will be questioned and documented in the electronic Case Report Form.
Technical feasibility: Percentage of not performed PVE | During the procedure of portal vein embolization
  Percutaneous access to the portal vein is achieved under general anesthesia with ultrasound or fluoroscopic control. Venous cartography of the liver is achieved with fluoroscopic control. PVE technique remains unchanged but a mixture of absorbable embolization agent is injected.
  Adverse events will be questioned and documented in the electronic Case Report Form.
Per and post procedure (within 6 weeks) morbidity | During PVE and within 6 weeks after embolization
  Portal thrombosis, pulmonary embolism and other complications
Liver tolerance | At Day0, Day1 and Day7 after portal vein embolization
  Liver function tests at Day0, Day1 and Day7 after portal vein embolization
Rate of portal partial and complete recanalization (subsegmental, segmental and sectorial) | 4-6 weeks after portal vein embolization
  During CT scan series performed 4 to 6 weeks after PVE, portal venous tree patency will be assessed by one independent blind observer.
Rate of patients considered after portal vein embolization for surgery in their centers | Through study completion, an average of 14 months
  All patients who underwent PVE procedure with sufficiently hypertrophy of non-embolized liver segments will return to hospital in order to undergo liver surgery. Decision to proceed with surgery will be left on investigator's discretion.
Rate of patients that finally undergo surgery | Through study completion, an average of 14 months
  All patients who underwent PVE procedure with sufficiently hypertrophy of non-embolized liver segments will return to hospital in order to undergo liver surgery. Decision to proceed with surgery will be left on investigator's discretion.
Inflammation and adhesions during portal pedicles dissection | During liver surgery.
  Assessment of the level of inflammation and adhesions will be performed during portal pedicles dissection. The senior surgeon will evaluate the level of inflammation and adhesions during portal pedicles dissection using a quantitative scale.
Intraoperative morbidity. | Up to 90 days following liver surgery.
  Liver failure and other complications due to surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Antoine Béclère, Clamart, France

IPD SHARING:
Plan to Share IPD: No